CLINICAL TRIAL: NCT03929419
Title: "Effect of Central Insulin Administration on Whole-body Insulin Sensitivity in Women"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 568/2018BO1
Record Dates: First submitted 2019-04-15; First posted 2019-04-26 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2020-11

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin nasal spray (Active Comparator): 160 Units of human insulin as nasal spray
  Interventions: Drug: intranasal insulin
- Placebo nasal spray (Placebo Comparator): Nasal spray containing placebo solution
  Interventions: Drug: Placebo spray

INTERVENTIONS:
Drug: intranasal insulin — application of 160 units human insulin
  Arms: Insulin nasal spray
Drug: Placebo spray — nasal spray containing placebo solution
  Arms: Placebo nasal spray

SUMMARY:
The human brain is an insulin sensitive organ. Brain insulin action modulates peripheral insulin sensitivity in young lean men. As a underlying mechanism, the investigators previously detected suppression of endogenous glucose production and stimulation of glucose disappearance to peripheral tissue in response to brain insulin delivery by nasal spray. Whether this holds true in young woman is unknown, since differences in brain insulin response between sexes have been reported. The investigators will address this question by combining the delivery of insulin to the brain as nasal spray with hyperinsulinemic euglycemic clamp experiments in natural cycling women.

In the planned randomized, placebo controlled cross-over study, female participants will undergo four hyperinsulinemic euglycemic experiments with tracer dilution, two in the first phase and two in the second phase of their menstrual cycle. On one of the study days per menstrual phase, subjects will receive intranasal insulin administration, on the other placebo spray. The protocol has been successfully applied previously in men. Based on the results of this trial, the investigators calculated a required sample size of N=10 for the planned study in women.

These experiments will help to better understand the role of brain insulin action in a broader sense. The results can be the basis for larger clinical trials that address the sex-specific impact of brain insulin resistance for glucose metabolism and diabetes risk.

DETAILED DESCRIPTION:
"Effect of central insulin administration on whole-body insulin sensitivity in women" The human brain is an insulin sensitive organ. Brain insulin action modulates peripheral insulin sensitivity in young lean men. As a underlying mechanism, the investigators previously detected suppression of endogenous glucose production and stimulation of glucose disappearance to peripheral tissue in response to brain insulin delivery by nasal spray. Whether this holds true in young woman is unknown, since differences in brain insulin response between sexes have been reported. The investigators will address this question by combining the delivery of insulin to the brain as nasal spray with hyperinsulinemic euglycemic clamp experiments in natural cycling women.

In the planned randomized, placebo controlled cross-over study, female participants will undergo four hyperinsulinemic euglycemic experiments with tracer dilution, two in the first phase and two in the second phase of their menstrual cycle. On one of the study days per menstrual phase, subjects will receive intranasal insulin administration, on the other placebo spray. The protocol has been successfully applied previously in men. Based on the results of this trial, the investigators calculated a required sample size of N=10 for the planned study in women.

These experiments will help to better understand the role of brain insulin action in a broader sense. The results can be the basis for larger clinical trials that address the sex-specific impact of brain insulin resistance for glucose metabolism and diabetes risk.

ELIGIBILITY:
Inclusion Criteria:

* female volunteer adults
* HbA1c <6.0%
* Age between 18 and 30 years
* Standard routine laboratory
* No underlying diseases
* No medication
* No hormonal contraception
* Understanding of the explanations of the study and the instructions

Exclusion Criteria:

* Persons with limited temperature perception and / or increased temperature Sensitivity to warming of the body
* Cardiovascular disease, such as manifest coronary Heart disease, heart failure greater than NYHA 2, recent myocardial infarction
* People with a hearing disorder or increased sensitivity to loud Sounds
* persons with claustrophobia
* Minors or non-consenting subjects are also excluded
* Pregnancy or breastfeeding women
* Surgery less than 3 months ago
* Simultaneous participation in other interventional studies
* Acute illness or infection within the last 4 weeks
* Neurological and psychiatric disorders
* Subjects with hemoglobin Hb <12g / dl (at screening)
* Allergic diseases
* Individuals with a history of heparin-induced thrombocytopenia (HIT)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2019-04-21 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in the peripheral insulin sensitivity | 60-90 minutes and 150-210 minutes during euglycemic clamp
  Effect of nasal insulin versus placebo on peripheral insulin sensitivity assessed by euglycemic hyperinsulinemic clamp.

SECONDARY OUTCOMES:
Correlation with autonomous nervous system activity | 70-80 minutes and 190-200 minutes during euglycemic clamp
  Correlation of the change in peripheral insulin sensitivity by central insulin action with the simultaneous change of the autonomous nervous system (measured by heart rate variability).
Differential effects dependent on female sexual hormones | 60-90 minutes and 150-210 minutes during euglycemic clamp
  Correlation of the change in peripheral insulin sensitivity by central insulin action dependent on the time point in menstrual cycle
Effect of menstrual cycle on insulin sensitivity before spray application | 60-90minutes
  Will be measured by hyperinsulinemic euglycemic clamp
Effect of menstrual cycle on brain insulin sensitivity | 60-90 minutes
  Brain insulin sensitivity will be assessed by functional magnetic resonance imaging combined with intranasal insulin administration during the follicular and the luteal phase of the menstrual cycle
Effect of menstrual cycle on processing of food cues in the brain | 20 minutes
  Processing of food cues in the brain will be assessed by functional magnetic resonance imaging during the follicular and the luteal phase of the menstrual cycle

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hummel J, Benkendorff C, Fritsche L, Prystupa K, Vosseler A, Gancheva S, Trenkamp S, Birkenfeld AL, Preissl H, Roden M, Haring HU, Fritsche A, Peter A, Wagner R, Kullmann S, Heni M. Brain insulin action on peripheral insulin sensitivity in women depends on menstrual cycle phase. Nat Metab. 2023 Sep;5(9):1475-1482. doi: 10.1038/s42255-023-00869-w. Epub 2023 Sep 21. PMID 37735274